CLINICAL TRIAL: NCT03184610
Title: Distinguishing Healthy and Keratoconic Eyes Using Ultrahigh-Resolution Optical Coherence Tomography (UHR-OCT) Based Corneal Epithelium Thickness Mapping
Brief Title: Distinguishing Healthy and Keratoconic Eyes Using Ultrahigh-Resolution OCT
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerald Schmidinger, Ass.Prof. PD Dr. Gerald Schmidinger, Medical University of Vienna
Other Study IDs: 1160/2014
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Keratoconus
Keywords: Keratoconus; Optical Coherence Tomography; Corneal Epithelium Thickness Maps
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OCT-scanning: Patients with Keratoconus are scanned with an OCT-Prototype
  Interventions: Device: OCT-scanning
- OCT-scanning for volunteers: Volunteers with healthy eyes are scanned with an OCT-Prototype
  Interventions: Device: OCT-scanning

INTERVENTIONS:
Device: OCT-scanning — All participants will be scanned with a OCT-device

SUMMARY:
The OCT used in this trial offers the advantage of both a non-contact method and a very high axial resolution. Determined parameters with the highest potential of diagnostic discrimination between eyes with Keratoconus and healthy eyes are investigated. Aim of this trial is to investigate differences of specific parameters of epithelium thickness maps at healthy eyes and eyes with Keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* Existence of Keratoconus
* written informed consent obtained

Exclusion Criteria:

* Earlier surgery such as PK, CXL, relaxing incisions
* Systemic diseases

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eyes with Keratoconus Healthy eyes
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Corneal Epithelium Thickness | One visit
  Parameters collected from epithelium thickness data and maps

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Ophthalmology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No